CLINICAL TRIAL: NCT05310240
Title: Evaluation of Prognostic Radiological Parameters on the Outcome After Hip Arthroscopy, a Cross-sectional Study
Brief Title: Analysis of the Relevance of Radiologic Parameters on the Outcome After Hip Arthroscopy
Status: Completed | Type: Observational
Sponsor: Bezirkskrankenhaus St. Johann in Tirol (Other)
Responsible Party: Principal Investigator, Moritz Wagner, Prinicpal investigator Dr. med. univ. Moritz Wagner, Bezirkskrankenhaus St. Johann in Tirol
Other Study IDs: 1199/2021
Record Dates: First submitted 2022-03-16; First posted 2022-04-04 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-08

CONDITIONS: Femoro-acetabular Impingement; Hip Impingement Syndrome; Hip Disease
Keywords: magnetic resonance arthrography; hip arthroscopy
MeSH Terms: conditions — Femoracetabular Impingement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hip arthroscopy: Patients that underwent hip arthroscopy at this department between 2013 and 2021.
  Interventions: Procedure: Hip arthroscopy

INTERVENTIONS:
Procedure: Hip arthroscopy — Arthroscopic surgery of the hip

SUMMARY:
Joint-preserving surgery with arthroscopic techniques of the hip follows detailed radiological assessment including plain radiography of the hips and magnetic resonance arthrography (MRI). The purpose of this study was to compare features on radiography and MRI of the hip before surgery and assess their prognostic value on the outcome after surgery.

DETAILED DESCRIPTION:
Hip arthroscopy is indicated for the treatment of a variety of pathologies of the hip, in patients without osteoarthritis. The diagnosis in patients with pain at the hip is made after history taking, clinical examination and radiological evaluation with plain radiography in a standardized technique and a magnetic resonance arthrography of the hip. The main indications for hip arthroscopy include CAM-type femoroacetabular impingement (FAI) necessitating bony decompression and chondro-labral tears necessitating arthroscopic repair or debridement. The purpose of this radiological non-interventional outcome study was to assess features on plain radiography and MRI in favor of good outcome after hip arthroscopy.

This department performed 810 hip arthroscopies in the years of 2013 till 2021. All of those patients underwent standardized radiological evaluation with radiography and MRI. Radiographical parameters are assessed by a resident with experience in musculo-sceletal radiology, intra- and inter-observer reliability has been assessed for each parameter. All arthroscopies have been performed by two experience senior orthopedic surgeons. Ethical board approval has been obtained to follow-up on those patients. Follow-up includes the patient-reported outcome assessment using the iHOT12 score and the modified Harris hip score. The clinical end-point is the time till total hip arthroplasty (THA), a registry analysis of the Tyrolean Arthroplasty registry (TAR) has been performed. Statistical analysis is performed using ANOVA and Fishers T-Tests, the level of significance is .05.

ELIGIBILITY:
Inclusion Criteria:

* Hip arthroscopy from 2013-2021 at this department.

Exclusion Criteria:

* Age below 18 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 810 patients received hip arthroscopy at this institution. All of those patients received an magnetic resonance arthrography.
Sampling Method: Non-Probability Sample
Enrollment: 810 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
prosthetic-free survival | Through study completion, an average of 1 year
  The number of days between hip arthroscopy and total hip arthroplasty. This parameter is assessed with the help of a joint-replacement registry for all subjects.

SECONDARY OUTCOMES:
iHOT12 Score | Through study completion, an average of 1 year
  Patient reported outcome measurement with validation for patients after hip arthroscopy
modified Harris-Hip score | Through study completion, an average of 1 year
  Patient reported outcome measurement with validation for failure of joint-preserving procedures

CONTACTS AND LOCATIONS:
Locations (1):
- BKH St. Johann in Tirol, Sankt Johann in Tirol, Tyrol, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ross JR, Larson CM, Bedi A. Indications for Hip Arthroscopy. Sports Health. 2017 Sep/Oct;9(5):402-413. doi: 10.1177/1941738117712675. Epub 2017 Jul 5. PMID 28678628
- [Background] McCarthy JC, Glassner PJ. Correlation of magnetic resonance arthrography with revision hip arthroscopy. Clin Orthop Relat Res. 2013 Dec;471(12):4006-11. doi: 10.1007/s11999-013-3202-5. Epub 2013 Aug 1. PMID 23904247
- [Derived] Wagner M, Lindtner RA, Schaller L, Schmaranzer F, Schmaranzer E, Vavron P, Endstrasser F, Brunner A. Hip arthroscopy with initial access to the peripheral compartment for femoroacetabular impingement: midterm results from a large-scale patient cohort. J Orthop Traumatol. 2024 May 24;25(1):29. doi: 10.1186/s10195-024-00770-6. PMID 38789896